CLINICAL TRIAL: NCT07128251
Title: A Single-Arm, Multicenter, Exploratory Clinical Study of Transarterial Chemoembolization (TACE) Combined With Iparomlimab and Tuvonralimab Injection and Bevacizumab Injection for the Treatment of Unresectable, Non-Metastatic Hepatocellular Carcinoma (HCC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Qilu Hospital of Shandong University (Other); Henan Provincial People's Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Shanxi Provincial Cancer Hospital (Unknown); Xi'an International Medical Center Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Lianxin Liu，PhD, professor, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025KY309
Record Dates: First submitted 2025-08-13; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC); Immunotherapy; PD-1; CTLA-4; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): TACE → Iparomlimab and Tuvonralimab Injection (QL1706) + Bevacizumab Injection (Q3W, 2 cycles). On-demand TACE therapy will be administered concurrently, with a maximum of 4 TACE sessions permitted.
  Interventions: Procedure: TACE treatment; Drug: Iparomlimab and Tuvonralimab Injection (QL1706); Drug: Bevacizumab

INTERVENTIONS:
Procedure: TACE treatment — TACE treatment (cTACE): On-demand TACE therapy will be administered, with a maximum of 4 TACE sessions permitted.
Drug: Iparomlimab and Tuvonralimab Injection (QL1706) — Iparomlimab and Tuvonralimab Injection (QL1706): 7.5 mg/kg, intravenous infusion, Day 1 of each cycle, Q3W.
Drug: Bevacizumab — Bevacizumab Injection: 15 mg/kg, intravenous infusion, Day 1 of each cycle, Q3W.

SUMMARY:
This is a single-arm, multicenter, exploratory clinical study designed to evaluate the efficacy and safety of TACE combined with Iparomlimab and Tuvonralimab Injection and Bevacizumab Injection in patients with unresectable, non-metastatic HCC. The primary endpoint is PFS as assessed by the investigator based on RECIST v1.1 criteria.

DETAILED DESCRIPTION:
This is a single-arm, multicenter, exploratory clinical study designed to evaluate the efficacy and safety of TACE combined with Iparomlimab and Tuvonralimab Injection and Bevacizumab Injection in patients with unresectable, non-metastatic HCC. The primary endpoint is PFS as assessed by the investigator based on RECIST v1.1 criteria.

After signing the informed consent form (ICF) and passing screening, subjects will undergo the first TACE procedure. Conventional TACE (cTACE) will be performed using lipiodol as the embolic agent and epirubicin as the chemotherapeutic agent. Study drug administration will commence at least 2 weeks after the first TACE: Iparomlimab and Tuvonralimab Injection [7.5 mg/kg, intravenous infusion, Day 1 (D1) of each cycle, every 21 days (Q3W)] combined with Bevacizumab Injection [15 mg/kg, intravenous infusion, D1, Q3W]. Each treatment cycle is 21 days (Q3W). On-demand TACE therapy will be administered concurrently, with a maximum of 4 TACE sessions permitted. The interval between consecutive TACE sessions must be at least 4 weeks. Bevacizumab Injection must be withheld for at least 2 days prior to any TACE procedure. Study drug administration must resume at least 2 weeks after any TACE procedure. Subjects must have fully recovered from TACE prior to receiving study drugs. Investigators may delay dosing based on toxicity recovery, but study drugs should be administered as soon as feasible once requirements are met.

Treatment will continue until the investigator assesses no further clinical benefit for the subject, the subject experiences intolerable toxicity, withdraws consent, or meets other protocol-specified criteria for treatment discontinuation (whichever occurs first).

Safety Visits: After enrollment, safety assessments will be performed 2 weeks (14 ± 3 days) after each TACE procedure and on D1 of each study drug cycle prior to drug administration. Subjects will continue safety assessments and survival follow-up after treatment completion.

Safety Reporting Period: Starts from the first TACE treatment and ends 90 days after the last dose of Iparomlimab and Tuvonralimab Injection [non-serious adverse events (AEs) unrelated to study drugs are collected only until 30 days after the last dose], or 30 days after the last dose of Bevacizumab Injection, or 30 days after the last TACE procedure, whichever is later.

Survival Follow-up: After the safety visit period, survival status and subsequent anti-tumor therapies will be collected every 12 weeks (±7 days) via clinical or telephone follow-up until subject death, loss to follow-up, sponsor study termination, or other study completion criteria are met (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and provide written informed consent.
2. Age 18-75 years, inclusive (male or female).
3. Histologically or cytologically confirmed HCC, or clinically diagnosed HCC according to the *Clinical Practice Guidelines for Primary Liver Cancer (2024 Edition)*.
4. Barcelona Clinic Liver Cancer (BCLC) Stage A, B, or C, not amenable to curative treatment (e.g., surgical resection, liver transplantation, or ablation).
5. At least one measurable lesion according to RECIST v1.1 criteria.
6. Suitable candidate for Transarterial Chemoembolization (TACE) with no known allergy or contraindication to iodized oil or epirubicin.
7. Child-Pugh Liver Function Class A.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
9. Life expectancy ≥ 3 months.
10. Adequate organ and bone marrow function.
11. If positive for Hepatitis B Virus (HBV) infection, HBV DNA must be < 2000 IU/mL (< 10,000 copies/mL if only copies/mL units available at the site) and the subject must be willing to receive continuous antiviral therapy throughout the study period. Subjects positive for Hepatitis C Virus (HCV) RNA must receive antiviral therapy according to clinical guidelines.
12. Subjects with esophageal/gastric varices must undergo evaluation and appropriate management prior to enrollment.
13. Women of childbearing potential (WOCBP): Must have a negative serum human chorionic gonadotropin (hCG) test within 7 days prior to initiation of study treatment; must be non-lactating; must agree to use highly effective contraception methods from signing informed consent until 120 days after the last dose of study treatment. A woman is considered of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (hysterectomy, bilateral salpingectomy/oophorectomy). Male subjects with female partners of childbearing potential: Must agree to use highly effective contraception methods from signing informed consent until 120 days after the last dose of study treatment; must agree to refrain from sperm donation. Male subjects with pregnant partners must use condoms; no additional contraception is required.

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, mixed hepatocellular cholangiocarcinoma, or cholangiocarcinoma; history of other active malignancies within 5 years or concurrently with HCC. Cured localized tumors (e.g., basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder carcinoma, carcinoma *in situ* of the prostate, cervix, or breast) are permitted.
2. Presence of Vp3 or Vp4 portal vein tumor thrombosis (PVTT), any grade of hepatic vein or inferior vena cava invasion; any grade of bile duct invasion. *Note: Vp1 or Vp2 PVTT is permitted.*
3. Presence of extrahepatic spread (EHS).
4. Intrahepatic lesion(s) with maximum diameter ≥ 10 cm, > 10 intrahepatic lesions, or intrahepatic tumor burden ≥ 70% of liver volume, per RECIST v1.1.
5. Prior systemic anti-cancer therapy for HCC, including molecular targeted agents, cytotoxic chemotherapy, immunotherapy (e.g., immune checkpoint inhibitors, immune checkpoint agonists, cellular therapies), or biologic therapy (e.g., cancer vaccines, cytokines, growth factors).
6. Prior locoregional therapy for HCC, including therapeutic TACE, transarterial embolization (TAE), hepatic arterial infusion chemotherapy (HAIC), transarterial radioembolization (TARE).

1) Prior curative surgery or ablation is permitted; one session of prophylactic TACE following curative resection is permitted.

2) Prior percutaneous ethanol injection (PEI) or radiotherapy with curative intent is permitted.

7. Prior or planned organ transplantation or allogeneic bone marrow transplantation.

8. Current interstitial lung disease (ILD)/pneumonitis, history of ILD/pneumonitis requiring steroid treatment, or other pulmonary conditions that may interfere with the detection or management of immune-mediated pneumonitis (e.g., pulmonary fibrosis, organizing pneumonia [e.g., bronchiolitis obliterans], pneumoconiosis, drug-induced pneumonitis, idiopathic pneumonitis, or active pneumonia evidenced by screening chest computed tomography [CT] scan). Prior radiation pneumonitis within the radiation field is permitted. Active tuberculosis.

9. Active autoimmune disease or history of autoimmune disease with potential for recurrence (e.g., autoimmune hepatitis, interstitial pneumonitis, uveitis, colitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; subjects with hypothyroidism stable on hormone replacement are eligible). Conditions not requiring systemic therapy (e.g., vitiligo, psoriasis, alopecia), controlled Type I diabetes on insulin, or childhood asthma in complete remission without adult intervention are permitted. Asthma requiring bronchodilator therapy is excluded.

10. Clinically significant ascites requiring therapeutic paracentesis or drainage (Child-Pugh score >2 for ascites; asymptomatic ascites detected only radiographically is permitted); uncontrolled or moderate/large pleural effusion or pericardial effusion.

11. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg based on ≥2 measurements) despite antihypertensive therapy; history of hypertensive crisis or hypertensive encephalopathy.

12. Clinically significant cardiac disease. 13. History of spontaneous rupture of hepatic tumor(s). 14. History of hepatic encephalopathy. 15. History or presence of central nervous system metastases. 16. Congenital or acquired immunodeficiency (e.g., HIV infection). 17. Thromboembolic event within 3 months prior to treatment (e.g., cerebrovascular accident [including transient ischemic attack, cerebral hemorrhage, cerebral infarction], deep vein thrombosis, pulmonary embolism).

18. History of gastrointestinal (GI) bleeding within 6 months prior to treatment or high risk of GI bleeding (e.g., high-risk or severe esophageal/gastric varices, active GI ulceration, persistent fecal occult blood positivity). *Note: If fecal occult blood positive at baseline, repeat test; if persistently positive, esophagogastroduodenoscopy [EGD] required; exclusion if EGD shows varices/lesions with bleeding risk.* 19. Abdominal fistula, GI perforation, intra-abdominal abscess, or bowel obstruction within 6 months prior to treatment.

20. Major surgical procedure within 4 weeks prior to treatment or anticipated during study; unhealed wound, ulcer, or fracture within 4 weeks prior to treatment.

21. Coagulopathy or bleeding diathesis (e.g., hemophilia); use of antiplatelet agents (e.g., aspirin >325 mg/day, dipyridamole, ticlopidine, clopidogrel, cilostazol) or anticoagulants (e.g., warfarin, low molecular weight heparin) within 10 days prior to treatment.

22. Significant vascular disease within 6 months prior to treatment (e.g., aortic aneurysm requiring surgical repair, recent peripheral arterial thrombosis).

23. Severe infection within 4 weeks prior to treatment (e.g., requiring hospitalization for infection, bacteremia, or severe pneumonia complications); therapeutic antibiotics administered orally or intravenously within 2 weeks prior to treatment (prophylactic antibiotics, e.g., for UTI or COPD prevention, are permitted).

24. Known hypersensitivity to the active substances or excipients of **Iparomlimab and Tuvonralimab Injection**, **Bevacizumab Injection**, or epirubicin; history of severe hypersensitivity to any other monoclonal antibody or anti-angiogenic targeted therapy.

25. Use of immunosuppressive agents or systemic corticosteroids (>10 mg/day prednisone or equivalent) for immunosuppressive purposes within 2 weeks prior to treatment.

26. Administration of live attenuated vaccines within 4 weeks prior to treatment or planned during Iparomlimab and Tuvonralimab Injection treatment or within 60 days after the last dose.

27. Treatment with any investigational agent within 4 weeks or 5 half-lives (whichever is longer) prior to treatment initiation.Subjects with any other condition deemed by the investigator to potentially affect study results or lead to premature study termination (e.g., alcoholism, drug abuse, other severe medical/psychiatric disorders requiring concomitant therapy, significant laboratory abnormalities, or familial/societal factors compromising subject safety).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as assessed by the Investigator according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | 2-year
  Defined as the time from initiation of study intervention to the first occurrence of either investigator-assessed (RECIST v1.1) radiographic disease progression or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6-month
  Proportion of subjects achieving Complete Response (CR) or Partial Response (PR) among all enrolled subjects (assessed by investigators per RECIST v1.1 and mRECIST).
Disease Control Rate (DCR) | 6-month
  Proportion of subjects achieving CR, PR, or Stable Disease (SD) among all enrolled subjects (assessed by investigators per RECIST v1.1 and mRECIST)
Overall Survival (OS) | 3-year
  Time from the start of therapy to death from any cause.
Adverse event (AE) | 3-year
  Adverse events (AEs), Serious Adverse events (SAEs), surgery related safety.

IPD SHARING:
Plan to Share IPD: No